CLINICAL TRIAL: NCT07357038
Title: A Real-world Prospective Observational Study on the Efficacy and Safety of L-AmB for br- IFD in Children and Adolescent Patients With Hematological Malignancies Receiving Triazoles or Echinocandins Prophylaxis
Brief Title: A Real-world Prospective Observational Study on the Efficacy and Safety of L-AmB(Liposomal Amphotericin B) for br- IFD(Breakthrough Invasive Fungal Disease) in Children and Adolescent Patients With Hematological Malignancies Receiving Triazoles or Echinocandins Prophylaxis
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: QTJC2024077
Record Dates: First submitted 2025-09-23; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-09

CONDITIONS: Fungal Disease
Keywords: malignant hematological diseases; breakthrough; invasive fungal disease; liposomal amphotericin B
MeSH Terms: conditions — Mycoses; Invasive Fungal Infections | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children and adolescent patients with hematological malignancies who have breakthrough IFD: children and adolescent patients with hematological malignancies who have breakthrough IFD after receiving triazoles or echinocandins prophylaxis
  Interventions: Drug: Patients received the Drug: liposomal amphotericin B（AmBisome） for treatment

INTERVENTIONS:
Drug: Patients received the Drug: liposomal amphotericin B（AmBisome） for treatment — 1. This is a single center, prospective ,single-arm and observational study.
  2. Patients who meet the inclusion and exclusion criteria receive liposomal amphotericin B (L-AmB)(AmBisome) for antifungal therapy.
  Regarding the combination therapy: During the research period, it is allowed to combine with other antifungal drugs in combination and accurately record them. Researchers determine it based on the severity of the underlying disease, the recovery of immune suppression, and clinical response.
  Regarding the sequential therapy: During the research period, it is allowed to accept sequential therapy with other antifungal drugs and accurately record them. Researchers determine it based on the severity of the underlying disease, the recovery of immune suppression, and clinical response.
  Regarding the surgical treatment: If the patient's condition permits, surgical treatment can be accepted and explained.
  Dosage: All medication doses are to be administered in accordance with the drug

SUMMARY:
The goal of this observational study is to evaluate the efficacy the favorable response rate and safety of L-AmB(liposomal amphotericin B) for the treatment of br-IFD(breakthrough invasive fungal disease) in Chinese children and adolescent patients with hematological malignancies receiving triazoles/echinocandins antifungal prophylaxis.

The main question it aims to answer is:

1. Whether the L-AmB have the same efficacy in the treatment of br-IFD in Chinese children and adolescent with hematological malignancies who are receiving triazoles or echinocandins antifungal prophylaxis as in adults(compared with historical data)
2. Whether L-AmB may have better renal safety in Chinese children and adolescent than in adults (compared with historical data).

Chinese children and adolescent with hematological malignancies will taking L-AmB as part of their regular medical care for br-IFD. The efficacy and safety data will be recorded.

DETAILED DESCRIPTION:
This is a single center, prospective, single-arm and observational study. Patients with breakthrough IFD in children and adolescent patients with hematological malignancies receiving triazoles or echinocandins prophylaxis who meet the inclusion and exclusion criteria receive liposomal amphotericin B (L-AmB)(AmBisome) for antifungal therapy. The efficacy and safety will be observed.

The response rate is assumed to be 67%, a sample size of 38 will produce a two-sided 95% confi dence interval for response rate with a width 0.3 (30%). With a 10% dropout consideration, 43 patients will need to be enrolled.

The research objective of this study is to: (a) Evaluate the efficacy and safety of L-AmB for the treatment of br-IFD in Chinese children and adolescent patients with hematological malignancies receiving triazoles/echinocandins prophylaxis.

(b) Identify baseline characteristic that may be associated with better response rates treated with L-AmB.

These research objectives will contribute to a comprehensive understanding of the roles of L-AmB in the treatment of breakthrough IFD in children and adolescent patients, and provide scientific evidence for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* The children and adolescent patients with hematological malignancy received echinocandin/triazole for antifungal prophylaxis and diagnosed with br-IFD.

  1. Age: from 1 month to 18 years old.
  2. Diagnosed patients with hematological malignancy.
  3. Received echinocandin/triazole for antifungal prophylaxis at least 7 days.
  4. Br-IFD is defined as a proven, probable, and possible IFD diagnosed at least 7 days after the start of primary antifungal prophylaxis and by 7 days from the end of primary antifungal prophylaxis. Definitions of proven, probable and possible IFD based on the EORTC/MSG 2020 criteria.
  5. ECOG-PS(Eastern Cooperative Oncology Group Performance Status): 0-2 points.
  6. There are no organ dysfunction restrictions during the screening period that limit the use of this protocol.
  7. The guardian understands the research and signs written informed consent form.

Exclusion Criteria:

* (a) Received AmB formulation for prophylaxis or treatment within the past 30 days.

  (b) Confirmed allergy/rapid onset severe allergic reaction/intolerance to L-AmB (c) Has a history of other tumors and has received any treatment for this tumor within the past 3 years (d) HIV, active hepatitis B and active hepatitis C virus or syphilis infection (e) Suffering from mental illness or other conditions that prevent cooperation with research, treatment, and monitoring requirements (f) Serum creatinine level 2 times the upper limit of normal; Liver transaminase or alkaline phosphatase levels 5 times the upper limit of normal, bilirubin levels 3 times the upper limit of normal (g) Researchers believe that patients who are not suitable for inclusion

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: breakthrough IFD in children and adolescent patients with hematological malignancies receiving triazoles or echinocandins prophylaxis
Sampling Method: Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
The favorable response rate . | The favorable response rate at the end of L-AmB therapy( an average of 2 weeks). The favorable response rate: proportion of patients achieving complete or partial remission.

SECONDARY OUTCOMES:
Safety data | Through study completion, an average of 14 days.
  Monitor and record any adverse reactions that occur during treatment, with adverse reaction names and grades recorded and evaluated according to NCI-CTCAE V 5.0(National Cancer Institute - Common Terminology Criteria for Adverse Events Version 5.0), including but not limited to the following indicators: clinical symptoms such as infusion reactions; Laboratory tests such as nephrotoxicity related indicators (creatinine, glomerular filtration rate), electrolytes (hypokalemia, hypomagnesemia), hepatotoxicity related indicators (alanine aminotransferase, aspartate aminotransferase, presidential bilirubin, direct bilirubin, indirect bilirubin), electrocardiogram, cardiac enzymes, etc

CONTACTS AND LOCATIONS:
Locations (1):
- National Clinical Research Center for Blood Diseases, Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No